CLINICAL TRIAL: NCT01195610
Title: A Six Month Randomized Controlled Dietary Intervention Study of the New Nordic Diet vs Average Danish Diet in Adults (18-65y) Using the Shop Model for Optimal Dietary Adherence
Brief Title: Dietary Intervention With Shop Model - SHOPUS
Acronym: SHOPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Thomas Meinert Larsen, Associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B 260
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Nordic Diet (Experimental): New Nordic Diet
  Interventions: Behavioral: Dietary intervention
- Average Danish Diet (Experimental): Average Danish Diet
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Instruction to diet for 6 month

SUMMARY:
The objective is to investigate whether New Nordic Diet (NND) versus Average Danish Diet (ADD) in adults (18-65 y) with central obesity and components of the metabolic syndrome can improve body weight loss and risk markers of the metabolic syndrome, type 2 diabetes and cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* abdominal obesity

Exclusion Criteria:

* BMI > 45, previous weight change

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in body weight (kg) | 26 weeks
  Change in body weight from randomization to end of intervention

SECONDARY OUTCOMES:
Change in body fat percentage | 26 weeks
  Change in body fat percentage (DEXA-scanning)
Dietary compliance | 26 weeks
  Level of dietary compliance
Changes in components of the metabolic syndrome | 26 weeks
  Changes in the number of components of the metabolic syndrome
Achievement of 5% weight loss | 26 weeks
  Achievement of 5% weight loss from randomization to end of intervention

OTHER OUTCOMES:
Change in gastrointestinal microbial composition | 26 weeks
  Diet specific changes in relative abundance of microbial bacteria
Microbial composition and association with Body weight change | 26 weeks
  Diet specific change in body weight according to relative abundance of microbial bacteria, e.g., baseline Prevotella/Bacteroides ratio [proxy for enterotypes])
Molecular regulation of glucose homeostasis | 26 weeks
  Diet specific molecular regulation in adipose and muscle tissue
Human salivary amylase gene copy number (AMY1 CN) and association with Body weight change [ Time Frame: 26 weeks ] | 26 weeks
  Diet specific change in body weight according to AMY1 CN

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meinert Larsen, PhD, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Background] Roager HM, Licht TR, Poulsen SK, Larsen TM, Bahl MI. Microbial enterotypes, inferred by the prevotella-to-bacteroides ratio, remained stable during a 6-month randomized controlled diet intervention with the new nordic diet. Appl Environ Microbiol. 2014 Feb;80(3):1142-9. doi: 10.1128/AEM.03549-13. Epub 2013 Dec 2. PMID 24296500
- [Background] Hjorth MF, Roager HM, Larsen TM, Poulsen SK, Licht TR, Bahl MI, Zohar Y, Astrup A. Pre-treatment microbial Prevotella-to-Bacteroides ratio, determines body fat loss success during a 6-month randomized controlled diet intervention. Int J Obes (Lond). 2018 Mar;42(3):580-583. doi: 10.1038/ijo.2017.220. Epub 2017 Sep 8. PMID 28883543
- [Background] Fritzen AM, Lundsgaard AM, Jordy AB, Poulsen SK, Stender S, Pilegaard H, Astrup A, Larsen TM, Wojtaszewski JF, Richter EA, Kiens B. New Nordic Diet-Induced Weight Loss Is Accompanied by Changes in Metabolism and AMPK Signaling in Adipose Tissue. J Clin Endocrinol Metab. 2015 Sep;100(9):3509-19. doi: 10.1210/jc.2015-2079. Epub 2015 Jun 30. PMID 26126206
- [Result] Poulsen SK, Crone C, Astrup A, Larsen TM. Long-term adherence to the New Nordic Diet and the effects on body weight, anthropometry and blood pressure: a 12-month follow-up study. Eur J Nutr. 2015 Feb;54(1):67-76. doi: 10.1007/s00394-014-0686-z. Epub 2014 Mar 25. PMID 24664189
- [Result] Poulsen SK, Due A, Jordy AB, Kiens B, Stark KD, Stender S, Holst C, Astrup A, Larsen TM. Health effect of the New Nordic Diet in adults with increased waist circumference: a 6-mo randomized controlled trial. Am J Clin Nutr. 2014 Jan;99(1):35-45. doi: 10.3945/ajcn.113.069393. Epub 2013 Nov 20. PMID 24257725
- [Derived] Hjorth MF, Christensen L, Larsen TM, Roager HM, Krych L, Kot W, Nielsen DS, Ritz C, Astrup A. Pretreatment Prevotella-to-Bacteroides ratio and salivary amylase gene copy number as prognostic markers for dietary weight loss. Am J Clin Nutr. 2020 May 1;111(5):1079-1086. doi: 10.1093/ajcn/nqaa007. PMID 32034403
- [Derived] Acar E, Gurdeniz G, Khakimov B, Savorani F, Korndal SK, Larsen TM, Engelsen SB, Astrup A, Dragsted LO. Biomarkers of Individual Foods, and Separation of Diets Using Untargeted LC-MS-based Plasma Metabolomics in a Randomized Controlled Trial. Mol Nutr Food Res. 2019 Jan;63(1):e1800215. doi: 10.1002/mnfr.201800215. Epub 2018 Aug 26. PMID 30094970
- [Derived] Hjorth MF, Ritz C, Blaak EE, Saris WH, Langin D, Poulsen SK, Larsen TM, Sorensen TI, Zohar Y, Astrup A. Pretreatment fasting plasma glucose and insulin modify dietary weight loss success: results from 3 randomized clinical trials. Am J Clin Nutr. 2017 Aug;106(2):499-505. doi: 10.3945/ajcn.117.155200. Epub 2017 Jul 5. PMID 28679551
- [Derived] Khakimov B, Poulsen SK, Savorani F, Acar E, Gurdeniz G, Larsen TM, Astrup A, Dragsted LO, Engelsen SB. New Nordic Diet versus Average Danish Diet: A Randomized Controlled Trial Revealed Healthy Long-Term Effects of the New Nordic Diet by GC-MS Blood Plasma Metabolomics. J Proteome Res. 2016 Jun 3;15(6):1939-54. doi: 10.1021/acs.jproteome.6b00109. Epub 2016 May 20. PMID 27146725